CLINICAL TRIAL: NCT01063634
Title: Comparison of a Plastic Stent Without Central Lumen With Self Expandable Metal Stents in Patients With Malignant Distal Biliary Obstruction. A Randomized, Controlled Trial
Brief Title: Comparison of a Plastic Stent Without Central Lumen With Self Expandable Metal Stents in Patients With Malignant Distal Biliary Obstruction
Acronym: VIADUCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kliniken Ludwigsburg-Bietigheim gGmbH (Other)
Collaborators: Klinikum Ludwigshafen (Other); Universitätsmedizin Mannheim (Other)
Responsible Party: Medizinische Klinik I, Prof. Dr. K. Caca, Klinikum Ludiwgsburg
Other Study IDs: VIADUCT
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: To Evaluate Patency of the Viaduct Stent in Comparison to Metal Stents
Keywords: malignant biliary obstruction; viaduct; self-expandable metal stents

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a non-inferiority randomized study to compare a plastic stent without central lumen (VIADUCT) with self-expandable metal stents for treatment of malignant obstruction of the common bile duct. It is a non-interventional study, a CE mark for the VIADUCT stent exists.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven malignant biliary stenosis
* signs of biliary obstruction
* informed consent

Exclusion Criteria:

* age under 18
* Operations like Roux-Y, biliodigestive Anastomosis, BII
* life expectancy less than 3 months
* Karnfosky index less than 60%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with malignant obstruction of the common bile duct
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Estimated); Study Completion 2012-01 (Estimated)

SECONDARY OUTCOMES:
time to stent obstruction | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Ludwigsburg, Ludwigsburg, Germany

REFERENCES:
- [Derived] Schmidt A, Riecken B, Rische S, Klinger C, Jakobs R, Bechtler M, Kahler G, Dormann A, Caca K. Wing-shaped plastic stents vs. self-expandable metal stents for palliative drainage of malignant distal biliary obstruction: a randomized multicenter study. Endoscopy. 2015 May;47(5):430-6. doi: 10.1055/s-0034-1391232. Epub 2015 Jan 15. PMID 25590188